CLINICAL TRIAL: NCT01340365
Title: Tai Chi, Physiologic Complexity, and Healthy Aging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter Wayne, Assistant Professor in Medicine, Harvard University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010P-000279
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Aquatic Therapy; Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other)
  Interventions: Behavioral: Tai Chi
- Tai Chi (Experimental): Individuals will take part in community-based Tai Chi classes twice a week for 6 months as well as practice Tai Chi outside of class twice a week for the same 6 month period.
  Interventions: Behavioral: Tai Chi Exercise

INTERVENTIONS:
Behavioral: Tai Chi Exercise — Practicing Tai Chi exercise 4 times a week for 6 months - twice in a classroom and twice independently
  Arms: Tai Chi
Behavioral: Tai Chi — Usual care, individuals attend testing sessions for 6 months with testing at times 0, 3, and 6 months. Individuals in Usual Care receive 3 months of Tai Chi at the study end.
  Arms: Usual Care

SUMMARY:
To evaluate the effects of Tai Chi-a mind-body exercise--on age-related loss of physiological complexity (using fractal and entropy based measures), and to understand the relationship between complexity, function and adaptability, we will conduct a two-arm prospective randomized clinical trial. Our overarching goal is to evaluate if six months of Tai Chi training, compared to a waitlist control receiving standard medical care, can enhance physiological complexity and adaptability in older Tai Chi-naïve adults. Secondary goals of the study are to characterize the relationship between complexity biomarkers, measures of function, and resilience. This pilot study will inform a future more definitive trial by providing information on recruitment and retention, compliance, dose-dependent effects, preliminary estimates of effect size, and the optimal biomarkers of complexity, function, and adaptive capacity.

DETAILED DESCRIPTION:
Specific Aim #1: To determine if 6 months of Tai Chi training can increase complexity, function, and adaptive capacity of multiple physiological systems in older healthy adults. Specific Aim #2: To determine the relationships between biomarkers of physiological complexity, conventional measures of function and adaptive capacity. Statistical regression models will be used to determine relationships, both at baseline and overtime, between a) complexity biomarkers and measures of physical and cognitive function, and b) complexity biomarkers and adaptive capacity. Elucidating these relationships will further inform the interpretation of complexity biomarkers and provide insights into underlying component mechanisms contributing to complex physiological dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-79
* Living within the Greater Boston area
* Willing to adhere to 6 month Tai Chi training protocol

Exclusion Criteria:

* Chronic medical conditions, including: cardiovascular disease (myocardial infarction, angina, atrial fibrillation, or presence of a pacemaker), stroke, respiratory disease requiring daily use of an inhaler, diabetes mellitus, malignancies, neurological conditions (e.g., seizure disorder, Parkinson's, peripheral neuropathy), or other neuromuscular or musculoskeletal (requiring chronic use of pain medication) disease
* Acute medical condition requiring hospitalization within the past 6 months
* Self-reported (current) smoking or alcohol/drug abuse
* Uncontrolled Hypertension (resting SBP > 160 or DBP > 100mm Hg)
* Abnormal heart rate (resting HR > 100 bpm; <50bpm)
* Abnormal ECG (supraventricular tachyarrhythmia, atrial fibrillation, significant ST wave abnormality, 2nd and 3rd degree heart block)
* Pregnancy
* Current use of prescription medications including cardio- or vaso-active drugs and medications that can affect autonomic function including Beta agonists and antagonists, drugs with anticholinergic properties (e.g. tricyclic antidepressants or anti psychotics), and cholinesterase inhibitor
* Self-reported inability to walk continuously for 15 minutes unassisted
* Regular Tai Chi practice within past 5 years
* Regular participation in physical exercise on average 4 or more times per week

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Heart rate complexity | 0, 3, and 6 months
  Beat-to-beat variation measured using ECG for a 30 minute during seated quiet resting
Change in Center of Pressure complexity | 0, 3 and 6 months
  Center of pressure (COP) dynamics during quiet standing with eyes open

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Wayne, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Beth Israel Deaconess Medical Center, Brookline, Massachusetts, United States

REFERENCES:
- [Derived] Wayne PM, Gow BJ, Hou F, Ma Y, Hausdorff JM, Lo J, Rist PM, Peng CK, Lipsitz LA, Novak V, Manor B. Tai Chi training's effect on lower extremity muscle co-contraction during single- and dual-task gait: Cross-sectional and randomized trial studies. PLoS One. 2021 Jan 22;16(1):e0242963. doi: 10.1371/journal.pone.0242963. eCollection 2021. PMID 33481829
- [Derived] Gow BJ, Hausdorff JM, Manor B, Lipsitz LA, Macklin EA, Bonato P, Novak V, Peng CK, Ahn AC, Wayne PM. Can Tai Chi training impact fractal stride time dynamics, an index of gait health, in older adults? Cross-sectional and randomized trial studies. PLoS One. 2017 Oct 11;12(10):e0186212. doi: 10.1371/journal.pone.0186212. eCollection 2017. PMID 29020106
- [Derived] Walsh JN, Manor B, Hausdorff J, Novak V, Lipsitz L, Gow B, Macklin EA, Peng CK, Wayne PM. Impact of Short- and Long-term Tai Chi Mind-Body Exercise Training on Cognitive Function in Healthy Adults: Results From a Hybrid Observational Study and Randomized Trial. Glob Adv Health Med. 2015 Jul;4(4):38-48. doi: 10.7453/gahmj.2015.058. PMID 26331103
- [Derived] Wayne PM, Gow BJ, Costa MD, Peng CK, Lipsitz LA, Hausdorff JM, Davis RB, Walsh JN, Lough M, Novak V, Yeh GY, Ahn AC, Macklin EA, Manor B. Complexity-Based Measures Inform Effects of Tai Chi Training on Standing Postural Control: Cross-Sectional and Randomized Trial Studies. PLoS One. 2014 Dec 10;9(12):e114731. doi: 10.1371/journal.pone.0114731. eCollection 2014. PMID 25494333